CLINICAL TRIAL: NCT02345642
Title: A Hemodynamic Comparison of Stationary and Portable Pneumatic Compression Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14064
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 Healthy Patients without THA (Active Comparator): The 10 test subjects of this study arm will be healthy volunteers of various ages that are willing to have the efficacy of pneumatic compression tested on them.
  Interventions: Device: ActiveCare+SFT Supine; Device: VenaFlow Elite Supine; Device: ActiveCare+SFT Standing; Device: VenaFlow Elite Standing
- 10 Patients with THA on Post-Op Day 2 (Experimental): The 10 test subjects of this study arm will be primary THR patients of Dr. Westrich that have undergone uncomplicated THR surgery in which they are allowed to be full weight bearing by or before post-op day 2.
  Interventions: Device: ActiveCare+SFT Supine; Device: VenaFlow Elite Supine; Device: ActiveCare+SFT Standing; Device: VenaFlow Elite Standing

INTERVENTIONS:
Device: ActiveCare+SFT Supine
  Other Names: Portable Pneumatic Compression Device Supine
Device: VenaFlow Elite Supine
  Other Names: Stationary Pneumatic Compression Device Supine
Device: ActiveCare+SFT Standing
  Other Names: Portable Pneumatic Compression Device Standing
Device: VenaFlow Elite Standing
  Other Names: Stationary Pneumatic Compression Device Standing

SUMMARY:
We are comparing two pneumatic compression devices, VenaFlow (stationary) and MCS (portable) in both the supine an standing position. We will start supine and will take 3 baseline measurements of venous velocity and then apply a device and take 3 measurements of the increase in peak venous velocity. We will repeat this with the second device. We will then have the subject stand and repeat the above with each device. We will randomize the order of the devices in the supine and standing position. This study will involve 10 healthy subjects of various ages and 10 total hip replacements (THR) patients.

ELIGIBILITY:
Inclusion Criteria:

Phase one: 10 healthy test subjects will be included of various ages. They will have each pneumatic compression device applied in the supine and then standing positions.

Phase two: 10 patients following THR on postoperative day #2 will be included. These patients will agree to participate in the study and have to be able to stand for approximately 10 minutes.

Exclusion Criteria:

* Patients with lymphedema
* Patients with peripheral vascular disease (chronic venous insufficiency)
* Patients who do not wish to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucian Warth, MD, Study Director — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Westrich GH, Specht LM, Sharrock NE, Windsor RE, Sculco TP, Haas SB, Trombley JF, Peterson M. Venous haemodynamics after total knee arthroplasty: evaluation of active dorsal to plantar flexion and several mechanical compression devices. J Bone Joint Surg Br. 1998 Nov;80(6):1057-66. doi: 10.1302/0301-620x.80b6.8627. PMID 9853503
- [Background] Westrich GH, Specht LM, Sharrock NE, Sculco TP, Salvati EA, Pellicci PM, Trombley JF, Peterson M. Pneumatic compression hemodynamics in total hip arthroplasty. Clin Orthop Relat Res. 2000 Mar;(372):180-91. doi: 10.1097/00003086-200003000-00020. PMID 10738427
- [Background] Johanson NA, Lachiewicz PF, Lieberman JR, Lotke PA, Parvizi J, Pellegrini V, Stringer TA, Tornetta P 3rd, Haralson RH 3rd, Watters WC 3rd. Prevention of symptomatic pulmonary embolism in patients undergoing total hip or knee arthroplasty. J Am Acad Orthop Surg. 2009 Mar;17(3):183-96. doi: 10.5435/00124635-200903000-00007. PMID 19264711
- [Background] Pitto RP, Hamer H, Heiss-Dunlop W, Kuehle J. Mechanical prophylaxis of deep-vein thrombosis after total hip replacement a randomised clinical trial. J Bone Joint Surg Br. 2004 Jul;86(5):639-42. doi: 10.1302/0301-620x.86b5.14763. PMID 15274256
- [Background] Ben-Galim P, Steinberg EL, Rosenblatt Y, Parnes N, Menahem A, Arbel R. A miniature and mobile intermittent pneumatic compression device for the prevention of deep-vein thrombosis after joint replacement. Acta Orthop Scand. 2004 Oct;75(5):584-7. doi: 10.1080/00016470410001466. PMID 15513491
- [Background] Froimson MI, Murray TG, Fazekas AF. Venous thromboembolic disease reduction with a portable pneumatic compression device. J Arthroplasty. 2009 Feb;24(2):310-6. doi: 10.1016/j.arth.2007.10.030. Epub 2008 Apr 8. PMID 18534456
- [Background] Murakami M, McDill TL, Cindrick-Pounds L, Loran DB, Woodside KJ, Mileski WJ, Hunter GC, Killewich LA. Deep venous thrombosis prophylaxis in trauma: improved compliance with a novel miniaturized pneumatic compression device. J Vasc Surg. 2003 Nov;38(5):923-7. doi: 10.1016/s0741-5214(03)00792-4. PMID 14603195
- [Background] Colwell CW Jr, Spiro TE, Trowbridge AA, Morris BA, Kwaan HC, Blaha JD, Comerota AJ, Skoutakis VA. Use of enoxaparin, a low-molecular-weight heparin, and unfractionated heparin for the prevention of deep venous thrombosis after elective hip replacement. A clinical trial comparing efficacy and safety. Enoxaparin Clinical Trial Group. J Bone Joint Surg Am. 1994 Jan;76(1):3-14. doi: 10.2106/00004623-199401000-00002. PMID 8288662
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Silbersack Y, Taute BM, Hein W, Podhaisky H. Prevention of deep-vein thrombosis after total hip and knee replacement. Low-molecular-weight heparin in combination with intermittent pneumatic compression. J Bone Joint Surg Br. 2004 Aug;86(6):809-12. doi: 10.1302/0301-620x.86b6.13958. PMID 15330019
- [Background] Edwards JZ, Pulido PA, Ezzet KA, Copp SN, Walker RH, Colwell CW Jr. Portable compression device and low-molecular-weight heparin compared with low-molecular-weight heparin for thromboprophylaxis after total joint arthroplasty. J Arthroplasty. 2008 Dec;23(8):1122-7. doi: 10.1016/j.arth.2007.11.006. Epub 2008 Apr 2. PMID 18534421
- See also: VenaFlow Elite Description on DJO Global's website — http://www.djoglobal.com/products/venaflow/venaflow-elite-system
- See also: ActiveCare+SVT Description on MCS's website — http://www.mcsmed.com/activecare_sft_2.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 Healthy Patients Without THA: The 10 test subjects of this study arm will be healthy volunteers of various ages that are willing to have the efficacy of pneumatic compression tested on them. A randomization technique was used to determine laterality and sequence of study events.
  ActiveCare+SFT Supine
  VenaFlow Elite Supine
  ActiveCare+SFT Standing
  VenaFlow Elite Standing
- 10 Patients With THA on Post-Op Day 2: The 10 test subjects of this study arm will be primary THR patients of Dr. Westrich that have undergone uncomplicated THR surgery in which they are allowed to be full weight bearing by or before post-op day 2.
  ActiveCare+SFT Supine
  VenaFlow Elite Supine
  ActiveCare+SFT Standing
  VenaFlow Elite Standing
Period: Overall Study
Arm/Group | 10 Healthy Patients Without THA | 10 Patients With THA on Post-Op Day 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 10 Healthy Patients Without THA: The 10 test subjects of this study arm will be healthy volunteers of various ages that are willing to have the efficacy of pneumatic compression tested on them.
  ActiveCare+SFT Supine
  VenaFlow Elite Supine
  ActiveCare+SFT Standing
  VenaFlow Elite Standing
- Total: Total of all reporting groups
Arm/Group | 10 Healthy Patients Without THA | 10 Patients With THA on Post-Op Day 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 5 | 5
Age, Continuous [Mean (Full Range); unit: years] | 28.7 [21 to 43] | 64.6 [55 to 70] | 46.65 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Peak Venous Velocity
Description: Ultrasound of the venous system just below the saphenofemoral junction to assess the venous velocity will be taken before and after application the VenaFlow and the ActiveCare+S.F.T pneumatic compression devices. Change from Baseline in Peak Venous Velocity 30 minutes after Device is applied is recorded.
Time Frame: Change from Baseline in Peak Venous Velocity 30 minutes after Device is Applied
Measure: Mean (Full Range); unit: cm/s
Arm/Group | 10 Healthy Patients Without THA | 10 Patients With THA on Post-Op Day 2
Number analyzed (Participants) | 10 | 10
cm/s
  Delta PVV from before to after Venaflow (Standing) | 127.9 [40 to 188] | 155.7 [106 to 270]
  Delta PVV from before to after Venaflow (Supine) | 87.1 [51 to 204] | 86.8 [26 to 165]
  delta PVV from before to after Activeca (Standing) | 32.6 [16 to 44] | 41.9 [11 to 85]
  delta PVV from before to after Activecare (supine) | 40.5 [9 to 66] | 37.8 [28 to 51]

ADVERSE EVENTS:
Arm/Group | 10 Healthy Patients Without THA | 10 Patients With THA on Post-Op Day 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No